CLINICAL TRIAL: NCT03848117
Title: Effects of Mulligan and Cyriax Approach in Patients With Subacute Lateral Epicondylitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Sammar Abbas, Physiotherapist, Isra University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIRS-1702-M.Phil OPT-006
Record Dates: First submitted 2019-01-26; First posted 2019-02-20 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Lateral Epicondylitis
Keywords: Patient Rated Tennis Elbow Evaluation (PRTEE); Mobilization with movement; Deep Transverse friction massage
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned into two groups: Cyriax Approach group and Mulligan approach group. A coin was flipped at start of data collection for the first patient to be assigned odd number and included in cyriax group. Later on odd and even numbered patients were included in specific group. Additionally, data was collected from lateral epicondylitis patients visiting the DHQ Hospital Bahawalnagar.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (DTF massage & Mill's manipulation)(Group 1) (Active Comparator): For any given subject in group 1, PRTEE pain and functional disability evaluations and Hand grip strength were completed on the same day. Then each subject in 1st group completed 4 weeks of physical therapy sessions which were aimed to decrease pain, increase functional activity level, and improve hand grip strength. Each subject was evaluated for changes in symptoms on 1st week, 2nd week, 3rd week and 4th week.
  Interventions: Other: Cyriax approach i.e. DTF massage and Mill's manipulation
- ( Taping & MWM) (Group 2). (Active Comparator): For any given subject in group 2, PRTEE pain and functional disability evaluations and Hand grip strength were completed on the same day. Then each subject in second group completed 4 weeks of physical therapy sessions which were aimed to decrease pain, increase functional activity level, and improve hand grip strength. Each subject was evaluated for changes in symptoms on 1st week, 2nd week, 3rd week and 4th week.
  Interventions: Other: Mulligan approach i.e. Taping and MWM

INTERVENTIONS:
Other: Cyriax approach i.e. DTF massage and Mill's manipulation — Each patient in group I i.e. Cyriax group was given 20-minute session. Each session started in sitting position and initially deep transverse friction massage was done at lateral compartment of the elbow joint and immediately after that mill's manipulation at elbow joint with flexion at wrist joint in pronated arm position. This session was repeated three times a week for one month (Total 12 sessions/ one month).
  Arms: (DTF massage & Mill's manipulation)(Group 1)
Other: Mulligan approach i.e. Taping and MWM — Each patient in group II i.e. Mulligan group was given 30 to 45-minute session. Each session started in sitting position and it included mobilization with movement which was given in such a way that initially lateral glide at elbow joint was performed and after holding it, I asked the patient to make a fist and open the fist. In this way, I repeated this procedure 36 times and after 12 repetitions, a short rest period was given. Taping was applied after mobilization around the elbow joint over extensor carpi radialis muscles. This session was repeated three times a week for one month (Total 12 sessions/ one month).
  Arms: ( Taping & MWM) (Group 2).

SUMMARY:
Lateral epicondylitis (LE) is a pain causing musculoskeletal disease which mainly occurs due to the over exertion or over use of extensors of wrist mainly ECRB and pain is felt at the origin of common extensor tendon. This study was focused to assess the effectiveness of cyriax approach and mulligan approach to improve the functional status of sub acute lateral epicondylitis patients through patient related tennis elbow evaluation form.

DETAILED DESCRIPTION:
A total of 39 athletes with knee pain were recruited and randomly divided into two groups. 30 subjects fulfilled the inclusion criteria and were part of this trial, 15 in each group.The data was collected through general demographic questionnaire, PRTEE questionnaire to determine the level of pain and functional disability and Hand grip strength chart to measure grip strength while having epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Age group 20-50 years of both gender.
* Vas < 7
* Positive mills test and cozens test.
* Local tenderness on palpation over lateral epicondyle of the humerus.
* From sub-acute to chronic more than 2 weeks.

Exclusion Criteria:

* Any previous pathology of bone around elbow.
* Corticosteroid injection in the preceeding 3 months.
* Absence of clinical signs of tennis elbow.
* Any other systemic illness like metabolic, metastatic, infective disorders.
* Any other neurological abnormalities.
* Allergies to Mulligan tape.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Patient related tennis elbow evaluation pain scale | Upto 4 weeks
  Pain associated with daily tasks is measured through Patient related tennis elbow evaluation pain scale with categories as "0" for no pain and "10" for worst imaginable pain.
Patient related tennis elbow evaluation functional disability scale | Upto 4 weeks
  Degree of difficulty in performing daily tasks associated with elbow joint is measured through Patient related tennis elbow evaluation functional disability scale in categories as "0" for no difficulty in task and "10" for unable to do a task.

SECONDARY OUTCOMES:
Hand grip strength chart index | Upto 4 weeks
  It is also measured through hand grip dynamo meter with reference values according to gender description.

CONTACTS AND LOCATIONS:
Locations (1):
- Sammar Abbas, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR